CLINICAL TRIAL: NCT07190807
Title: Managing Pain Using Optimized Sequences by Adjusting Parameters With Independent Current Control (MOSAIC Study)
Brief Title: Managing Pain Using Optimized Sequences by Adjusting Parameters With Independent Current Control
Acronym: MOSAIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4116
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain; Intractable Pain; Low Back Pain; Chronic Low-back Pain; Chronic Leg Pain; Leg Pain
Keywords: Spinal Cord Stimulation
MeSH Terms: conditions — Chronic Pain; Pain, Intractable; Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Time Varied Pulse (TVP)-SCS settings (Experimental)
  Interventions: Device: Boston Scientific WaveWriter Alpha™ SCS Systems

INTERVENTIONS:
Device: Boston Scientific WaveWriter Alpha™ SCS Systems — Time Varied Pulse (TVP)-SCS settings

SUMMARY:
Study to evaluate the effectiveness of time variant pulse (TVP)-SCS in patients with chronic pain using commercially approved Boston Scientific SCS Systems per local Instructions for use (IFU).

In addition, to compile real-world clinical outcomes in subjects with chronic, intractable low back and/or leg pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Persistent spinal pain syndrome (PSPS) Type I (or non-surgical refractory back pain), or PSPS Type II (Failed Back Surgery Syndrome, FBSS) diagnosis.
* Diagnosed with chronic pain of the trunk and/or limbs for at least 6 months.
* 18 years of age or older when written informed consent is obtained
* Able to independently read and complete all questionnaires and assessments provided in English.
* Signed a valid, IRB or EC approved informed consent form (ICF) provided in English.

Key Exclusion Criteria:

* Any pain-related diagnosis, medical or psychological condition that, in the Investigator's judgment might confound reporting of study outcomes (e.g., vascular or neurogenic claudication, osteoarthritis, plantar fasciitis, pelvic pain, anginal pain, chronic migraine, acute herniated disc, malignancy, untreated major depression, injury claim).
* Significant cognitive impairment at Screening and Baseline visit that, in the opinion of the Investigator, would reasonably be expected to impair the study candidate's ability to participate in the study
* A female who is pregnant, lactating, or is of childbearing potential and planning to get pregnant during the study or not using adequate contraception.
* Participating (or intends to participate) in another drug or device clinical trial that may influence the data that will be collected for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Targeted Pain Responder Rate | 3 months post-activation
  Proportion of subjects with 50% or greater reduction from Baseline Visit in average targeted pain intensity at 3 months post-activation

CONTACTS AND LOCATIONS:
Overall Officials: Natalie M Bloom Lyons, Study Director — Boston Scientific Corporation
Locations (7):
- United States (7):
  - Denver Back Pain Specialists, Greenwood, Colorado
  - Orlando Health Neuroscience Institute, Clermont, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Montefiore Medical Center, The Bronx, New York
  - Fox Chase Pain Management, Trevose, Pennsylvania
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - Institute of Precision Pain Medicine, Corpus Christi, Texas